CLINICAL TRIAL: NCT06426641
Title: Polyethylene Wear Particle Analysis of Total Knee Arthroplasty -International Multicenter Study-
Brief Title: Polyethylene Wear Particle Analysis of TKA
Status: Active, not recruiting | Type: Observational
Sponsor: Osaka Metropolitan University (Other)
Collaborators: Mayo Clinic (Other); Istituto Ortopedico Rizzoli (Other); Hospital for Special Surgery, New York (Other)
Responsible Party: Principal Investigator, Yukihide Minoda, Associate professor, Osaka Metropolitan University
Other Study IDs: OMU 2023-108
Record Dates: First submitted 2024-05-16; First posted 2024-05-23 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Wear of Articular Bearing Surface of Prosthetic Joint; Total Knee Arthroplasty
Keywords: Polyethylene wear particle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — pericapsular tissue, which is removed during surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- polyethylene containing Vitamin E: polyethylene containing Vitamin E
  Interventions: Device: Polyethylene
- conventional polyethylene (no highly cross-linking): conventional polyethylene (no highly cross-linking)
  Interventions: Device: Polyethylene
- conventional polyethylene (with highly cross-linking): conventional polyethylene (with highly cross-linking)
  Interventions: Device: Polyethylene

INTERVENTIONS:
Device: Polyethylene — There is no intervention

SUMMARY:
The purpose of this study was to investigate whether polyethylene (Vitamin E-containing polyethylene), which has been newly introduced and widely used clinically as a biomaterial for tibial inserts in total knee arthroplasty, but whose mid- to long-term clinical results are still unknown, is more effective than conventional polyethylene.

Our goal is to clarify through an international multi-center joint study using in vivo polyethylene wear particle analysis, which the investigators developed as a method to provide early feedback, as to whether polyethylene wear debris production in vivo can be reduced.

DETAILED DESCRIPTION:
Anticipated medical contribution and significance In this study, the investigators investigate whether a newly introduced polyethylene (highly cross-linked polyethylene, vitamin E-containing polyethylene in vivo) can suppress wear debris production more than conventional polyethylene. If the newly introduced polyethylene can reduce wear debris production, it is expected to reduce failure of artificial joints in the future. However, if newly introduced polyethylene is actually increasing wear debris production, it could be an early alarm bell for surgeons around the world. In other words, the international and social impact of this research is extremely large.

Two unique requirements are necessary to carry out this research. Firstly, in vivo analysis of polyethylene wear particles is possible, and secondly, the number of surgical cases of revision knee arthroplasty targeted for investigation is large. The first requirement is that the applicants have published many English-language papers on in vivo polyethylene wear debris analysis, and that their facilities are the most suitable and fully capable of carrying out the analysis worldwide. be. The second requirement is that the investigators need to collaborate not only with our hospital but also with facilities that perform a large number of revision knee arthroplasty surgeries. Not only our hospital, but also our affiliated hospital, which is one of the facilities in Japan that performs the most knee joint surgeries (Naniwa Ikuno Hospital), and the hospital that performs the most knee joint surgeries worldwide (Mayo Clinic [USA]). , Hospital for Special Surgery [USA], Istituto Ortopedico Rizzoli [Italy]).

Research method In this study, the investigators conducted the following steps to determine the in vivo wear particles (number, size, and morphology) of conventional polyethylene, whose long-term results have already been clarified, and vitamin E-containing polyethylene, whose mid- to long-term results have not yet been clarified. Clarifying the difference [Figure 3].

Target of this research In this study, the investigators will focus on patients undergoing revision knee arthroplasty as a routine medical treatment.

First total joint replacement

* 30 patients using polyethylene containing Vitamin E
* 30 patients using conventional polyethylene (no highly cross-linking)
* 30 patients using conventional polyethylene (with highly cross-linking)

Accumulation of periarticular tissue In this study, the investigators will focus on patients undergoing revision knee arthroplasty as a routine medical treatment.

The test will be conducted after obtaining approval from the ethics committee at each facility and obtaining informed consent. The pericapsular tissue, which is removed during surgery and usually discarded, is obtained and fixed in formalin fixative. The tissue will be transported to the Department of Orthopedic Surgery, Osaka Public University Graduate School of Medicine for analysis. International transportation of tissues requires outsourcing to specialized companies with experience in transporting tissues from overseas.

Isolation of polyethylene wear debris The collected tissue around the joint capsule is immersed in 5M NaOH at 65°C for 1 hour to decompose the protein. Make a sucrose layer (5, 10, 20%) in a 14ml tube (14PA tube, Hitachi Koki Co, Ltd, Tokyo, Japan), add the dissolved solution, and place in an ultracentrifuge (CP100a, P28S1014 rotor, Hitachi Koki). Ultracentrifuge at 28,000 rpm [103,7009g] for 3 hours at 4°C. Prepare an isopropanol layer (0.90 and 0.96 g/mL) in a 40 ml tube (40PA tube, Hitachi Koki Co, Ltd, Tokyo, Japan), add the upper layer of sucrose layer, and centrifuge at 28,000 rpm (103,7009 g ) and perform ultracentrifugation at 4°C for 1 hour. The isopropanol interlayer is collected to isolate polyethylene wear debris.

Analysis of polyethylene wear debris The isopropanol interlayer is filtered through a 0.1 μm polycarbonate filter (VCTP 013-00, Millipore Corporation, Bedford, MA). Dry the polycarbonate filter, fix it on an aluminum pedestal (M4, Nisshin EM Co, Ltd, Tokyo, Japan), and apply platinum coating (E-1030 ion sputter, Hitachi Science Systems Ltd, Tokyo, Japan). Observe the polyethylene wear particles on the polycarbonate filter using a scanning electron microscope (S4700SI, Hitachi Ltd, Tokyo, Japan), and analyze the following items using an image analyzer (Mac Scope, Mitani Co, Tokyo, Japan).

* Number of polyethylene wear particles (number per 1g of tissue)
* Size (Equivalent circle diameter [μm])
* Shape (aspect ratio, roundness)

Comparison of iv vivo polyethylene wear powder morphology depending on polyethylene material The number, size, and form of polyethylene wear debris will be compared between conventional polyethylene, whose long-term results have already been clarified, and vitamin E-containing polyethylene, whose medium- to long-term results have not yet been clarified.

The investigators also investigated factors that affect polyethylene wear in vivo (age, height, weight, period from initial surgery to revision surgery, knee joint range of motion, knee prosthesis clinical score [Knee Society Score, University of California at Los Angeles activity score]).

Evaluation items (outcome) Main evaluation items: Polyethylene wear particle morphology (number of wear particles, equivalent circle diameter [㎛], aspect ratio, roundness) [Reason for setting primary endpoints] Because it is a standard evaluation item for evaluating polyethylene wear debris.

Secondary endpoints:

* Body mass index
* Knee joint range of motion
* Clinical score (2011Knee Society Score, Knee injury and Osteoarthritis Outcome Score for Joint Replacement, University of California at Los Angeles activity score) [Reason for setting secondary endpoints] Because it may affect the production of polyethylene wear debris.

Planned number of research subjects and basis for setting it (including cases where the number of research subjects is set without relying on statistical grounds) Total 90 cases

* 30 patients using polyethylene containing Vitamin E
* 30 patients using conventional polyethylene (no high cross-linking)
* 30 patients using conventional polyethylene (with high cross-linking) Rationale for setting: The target number of cases was determined from the number of cases at related institutions within the study period.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing revision knee arthroplasty within the study period
2. Patients over 20 years old
3. Patients who have received a sufficient explanation, have sufficient understanding, and have given their free written consent.
4. Patients who have passed 2 years or more since their first total knee arthroplasty

Exclusion Criteria:

1. Patients who are judged to be unsuitable as research subjects by the research physician

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing revision surgery
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-12-05 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of polyethylene wear particles | Time of revision surgery
  counts / g (tissue sample)
Equivalent circle diameter of polyethylene wear particles | Time of revision surgery
  Equivalent circle diameter (㎛)
Aspect ratio of polyethylene wear particles | Time of revision surgery
  Aspect ratio
Roundness of polyethylene wear particles | Time of revision surgery
  Roundness

SECONDARY OUTCOMES:
Body mass index | Time of revision surgery
  kg/m2
Knee joint extension angle | Time of revision surgery
  degrees
Knee joint flexion angle | Time of revision surgery
  degrees
2011 Knee Society Score: An "Objective" Knee Score | Time of revision surgery
  0(worse)-100(best)
2011 Knee Society Score: A Patient Satisfaction Score | Time of revision surgery
  0(worse)-40(best)
2011 Knee Society Score: A Patient Expectation Score | Time of revision surgery
  0(worse)-15(best)
2011 Knee Society Score: A Functional Activity Score | Time of revision surgery
  0(worse)-100(best)
Knee injury and Osteoarthritis Outcome Score for Joint Replacement | Time of revision surgery
  0(worse)-100(best)
University of California at Los Angeles activity score | Time of revision surgery
  1(worse)-10(best)

CONTACTS AND LOCATIONS:
Overall Officials: Yukihide Minoda, MD, PhD, Principal Investigator — Osaka Metropolitan University
Locations (2):
- Mayo Clinic, Rochester, Minnesota, United States
- Osaka Metroplitan Univerity, Osaka, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Minoda Y, Kobayashi A, Iwaki H, Iwakiri K, Inori F, Sugama R, Ikebuchi M, Kadoya Y, Takaoka K. In vivo analysis of polyethylene wear particles after total knee arthroplasty: the influence of improved materials and designs. J Bone Joint Surg Am. 2009 Nov;91 Suppl 6:67-73. doi: 10.2106/JBJS.I.00447. No abstract available. PMID 19884413
- [Result] Minoda Y, Kobayashi A, Iwaki H, Miyaguchi M, Kadoya Y, Ohashi H, Yamano Y, Takaoka K. Polyethylene wear particles in synovial fluid after total knee arthroplasty. Clin Orthop Relat Res. 2003 May;(410):165-72. doi: 10.1097/01.blo.0000063122.39522.c2. PMID 12771827